CLINICAL TRIAL: NCT03736434
Title: Brain Connections, Self-care and Blood Pressure in Black and African Americans With Problems With Memory
Brief Title: Brain Connections and Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kathy D. Wright, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2018H0136
Record Dates: First submitted 2018-11-07; First posted 2018-11-09 (Actual); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Hypertension; Mild Cognitive Impairment
Keywords: Mindfulness; Blood pressure; Hypertension; Mild Cognitive impairment (MCI); functional Magnetic resonance Imaging (fMRI); Hair cortisol
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Three aim randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Data collectors masked as to the hypotheses of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness plus DASH group (Experimental): Receives Mindfulness and DASH Diet education once a week for 8 weeks (2.5-hour sessions)
  Interventions: Behavioral: Mindfulness and DASH Diet Education; Behavioral: Education group
- Education Group (Active Comparator): The sham intervention includes general education on non-health related topics such as fire-safety and learning how to dispose of medication properly, once a week for 8 weeks (2.5-hour sessions)
  Interventions: Behavioral: Mindfulness and DASH Diet Education; Behavioral: Education group
- Control Group (No Intervention): Continue care as usual without intervention.

INTERVENTIONS:
Behavioral: Mindfulness and DASH Diet Education — Mindfulness and DASH diet education will include a didactic presentation on stress, theoretical material related to mindfulness, the somatic mind/body connection, relaxation, yoga, meditation, self-awareness, and bodily cues relating to emotional reactivity. Practices will include the body scan, gentle yoga movement, walking/sitting meditation, breathing, relaxation. Additionally, daily 20 min individual practices are done at least 5x/week delivered via a compact disc player or on a preloaded device. Each participant is asked to track his/her daily meditation practice and given a diary for adherence records. A combination of didactic, experiential, and "hands-on" activities will be done to deliver DASH diet guidelines.
  Arms: Education Group; Mindfulness plus DASH group
Behavioral: Education group — The attention control group will attend eight, 2.5 hours sessions on non-health topics such as personal safety, fire prevention, cold weather protection, disaster preparation, internet safety, aging in place, how to know when it's time to move and managing your money.
  Arms: Education Group; Mindfulness plus DASH group

SUMMARY:
This pilot randomized controlled study evaluates Mindfulness and DASH Diet resting state network and blood pressure in 36 (n=12 intervention; n=12 attention control; n = 12 control) Black and African American older adults with early Alzheimer's disease and related dementia disorders and hypertension.

DETAILED DESCRIPTION:
The purpose of this pilot randomized controlled study is to adapt a previously tested intervention to improve resting state network and blood pressure in 36 (n=12 intervention; n=12 attention control; n = 12 control) Black and African American older adults with early Alzheimer's disease and related dementia disorders and hypertension.

The study aims are to:

A.1. Establish the feasibility and acceptability of the intervention in Black and African Americans with Alzheimer's disease and related dementia disorders and hypertension.

H1: The intervention will be feasible and acceptable to Black and African Americans with Alzheimer's disease and related dementia disorders. Feasibility will be measured by recruitment, attendance, and attrition. Acceptability will be measured by a garnering feedback in a debriefing after each session.

A.2. Determine the effect size of the difference between the intervention, attention control, and control groups in resting state network connectivity and working memory and blood pressure to inform the sample size for the R01 trial.

H2: We hypothesize that compared to both control groups; the intervention group will have greater improvement in process measures of self-management mechanisms (self-efficacy, self-regulation, and emotion regulation), chronic stress, diet, and physical activity. The functional magnetic resonance imaging and blood pressure will be obtained at baseline and 3 months. The intervention group (Mindfulness + DASH) will have improved resting state network connectivity and blood pressure as compared to the attention control (2-hour group social time and brief lecture on a non-diet/mindfulness topic such as personal safety, fire safety, and disaster preparedness) and the control group (care as usual with no intervention). The Center for Cognitive and Behavioral Brain Imaging, Arts & Sciences co-investigators will analyze imaging data using their newly published statistical network model to quantify the subnetwork structures of the resting state network and evaluate changes of their topological properties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension with or without medication use
* Diagnosis of Alzheimer's disease or related dementia disorder or, if no formal diagnosis of Alzheimer's disease, then a Self-Assessment Gerocognitive Evaluation score 17-10 or a Montreal Cognitive Assessment Screen 25-19

Exclusion Criteria:

* Unable to understand spoken English
* Expect to move out of the area within six months
* fMRI imaging contraindicated (history of shrapnel, metal in the body, heart pacemaker, heart defibrillator, metal in the eye, gunshot wound, or some types of metal elsewhere within the body such as certain surgical clips for aneurysms in the head, heart valve prostheses, electrodes, and some other implanted devices) or claustrophobia. However, the participant can be included in the study without fMRI.
* Self-reported history of a stroke
* <6 on the Brief Assessment of Understanding of the Study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy D Wright, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited (August 2018-August 2019) from area clinics and the local African American Churches, The Charitable Pharmacy of Central Ohio. Additionally, participants will be recruited from the college of nursing Total Health and Wellness Center, local senior centers that service the African American community.
Pre-assignment Details: No participants were excluded. The participants were randomized into groups MIM DASH, non-hypertensive edcuation attention only, or true control. Unit of analysis is participants, not groups.
Period: Overall Study
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Started | 13 | 13 | 12
Completed | 12 | 13 | 6
Not Completed | 1 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group | Total
Number analyzed (Participants) | 13 | 13 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (5.9) | 71.9 (3.9) | 70.8 (5.5) | 72.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 10 | 31
  Male | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 13 | 12 | 38
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 12 | 38
Self-Administered Gerocognitive Examination (SAGE) [Mean (Standard Deviation); unit: units on a scale] — Self-Administered Gerocognitive Examination (SAGE), specifically designed to screen for mild cognitive impairment and early dementia. SAGE covers cognitive domains of orientation, language, memory, executive function, calculations, abstraction, and visuospatial abilities. The psychometric properties have been well validated with a 0.84 Spearman rank correlation between SAGE and a 1-day neuropsychiatric battery. Scores range from 0-22, score of 17 opr above is considered normal. Therefore higher scores indicate better outcomes.
  units on a scale | 13.3 (3.5) | 14.1 (2.6) | 13.4 (3.8) | 13.6 (3.3)
Number of chronic conditions [Mean (Standard Deviation); unit: Chronic Conditions] | 5 (1.3) | 4.5 (1.8) | 4.1 (1.0) | 4.8 (1.4)
Number of hypertension medications [Mean (Standard Deviation); unit: Number of medications] — Total number of medications participant is prescribed for hypertension
  Number of medications | 2.1 (0.9) | 1.9 (1.2) | 1.8 (1.0) | 2.0 (1.1)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 133.6 (14.4) | 140.4 (28.3) | 139.6 (12.8) | 137.8 (19.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 75.6 (9.6) | 78.3 (12.1) | 76.3 (13.3) | 76 (11.5)
Dietary Approaches to Stop Hypertension Questionnaire (DASH-Q) [Mean (Standard Deviation); unit: score on a scale] — DASH Q has 11 items focused on the consumption of DASH foods (e.g., fruits, nuts, and vegetables) in the past 7 days (Cronbach α = .83). The reference range for the DASH Q was 0-105 with higher scores indicating greater adherence to DASH diet.
  score on a scale | 70.0 (12.0) | 58.1 (11.1) | 69.1 (8.3) | 63.6 (12.6)
Cognitive and Affective Mindfulness Scale (Mindful Affect) [Mean (Standard Deviation); unit: score on a scale] — The Cognitive and Affective Mindfulness Scale (Cronbach α = .77)17 has 12 questions (reference range 0-48, higher scores indicate greater mindfulness affect) on a Likert scale regarding daily experiences such as "I rush through activities without being really attentive to them."
  score on a scale | 32.1 (5.9) | 33.7 (6.3) | 31.2 (6.0) | 31.2 (6.6)
Perceived Stress Scale [Mean (Standard Deviation); unit: score on a scale] — The Perceived Stress Scale has 10-items reference range 0-30 regarding stress over the past month (Cronbach α = 0.83).The cut point for moderate to high stress is 12 or more for persons aged 65 and older.
  score on a scale | 10.5 (7.1) | 9.7 (6.1) | 16.1 (10.1) | 12 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting State Network
Description: functional magnetic resonance imaging scans of brains utilizing and working memory test will be employed to measure change in resting state network
Time Frame: Baseline and 3 months
Population: This data point was unable to be collected, not able to complete MRIs.
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change in Systolic Blood Pressure
Description: Omron automatic blood pressure machine with small and large cuff sizes will be used to obtain blood pressure readings
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 13 | 13 | 12
mmHg | -10.4 (13.3) | -3.2 (17.4) | -13.8 (9.9)

3. Primary Outcome: Change in Diastolic Blood Pressure
Description: Omron automatic blood pressure machine with small and large cuff sizes will be used to obtain blood pressure readings
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 13 | 13 | 12
mmHg | -4.1 (7.9) | -3.4 (8.5) | -5.7 (6.1)

4. Secondary Outcome: Dietary Approaches to Stop Hypertension Questionnaire (DASH-Q) Change
Description: DASH Q has 11 items focused on the consumption of DASH foods (e.g., fruits, nuts, and vegetables) in the past 7 days (Cronbach α = .83). The reference range for the DASH Q was 0-105 with higher scores indicating greater adherence to DASH diet.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 13 | 13 | 12
score on a scale | -1.6 (10.8) | 0.2 (4.2) | -6 (9.3)

5. Secondary Outcome: Cognitive and Affective Mindfulness Scale Change
Description: The Cognitive and Affective Mindfulness Scale (Cronbach α = .77)17 has 12 questions (reference range 0-48, higher scores indicate greater mindfulness affect) on a Likert scale regarding daily experiences such as "I rush through activities without being really attentive to them."
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 13 | 13 | 12
score on a scale | -3.1 (9.1) | -2.1 (5.8) | 3.9 (5.7)

6. Secondary Outcome: Perceived Stress Scale Change
Description: The Perceived Stress Scale has 10-items reference range 0-30 regarding stress over the past month (Cronbach α = 0.83).1The cut point for moderate to high stress is 12 or more for persons aged 65 and older.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
Number analyzed (Participants) | 13 | 13 | 12
score on a scale | 1.2 (4.9) | 0.8 (7.4) | -5.9 (3.1)

ADVERSE EVENTS:
Time Frame: 3 months post intervention
Arm/Group | Mindfulness Plus DASH Group | Education Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT03736434/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT03736434/ICF_001.pdf